CLINICAL TRIAL: NCT07136597
Title: Investigating the Utility and Efficacy of Narrative Medicine Based Flash-writing on Healthcare Occupational Burnout and Stress Mitigation Among Atrium Health Wake Forest Baptist Faculty
Brief Title: Narrative Medicine Effects on Burnout and Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00126610
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-08

CONDITIONS: Healthcare Professionals
Keywords: stress mitigation; exhaustion; mental health challenges

STUDY DESIGN:
Intervention Model Description: narrative medicine based flash writing with burnout levels and stress response using a series of surveys and in-person workshops.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- narrative medicine workshops (Experimental): participants will be asked to attend 3/6 monthly narrative medicine workshops through the study's duration following an initial workshop that will be used to introduce the concepts of narrative medicine and flash writing
  Interventions: Behavioral: Narrative Medicine Workshop

INTERVENTIONS:
Behavioral: Narrative Medicine Workshop — participants will be asked to attend 3/6 monthly narrative medicine workshops through the study's duration following an initial workshop that will be used to introduce the concepts of narrative medicine and flash writing.
  Other Names: narrative medicine based flash-writing

SUMMARY:
A rising area of interest over the past several years has been on the issue of physician burnout. Burnout can be defined as a chronic occupational stress response characterized by multi-dimensional exhaustion and diminished sense of fulfillment in one's personal and professional life. Regarding the effects of emotional, occupational and physical stress on job satisfaction, standard of care and staff retention, it is important to determine meaningful methods to alleviate and prevent burnout among healthcare professionals.

DETAILED DESCRIPTION:
Common coping strategies for burnout and occupational stress are related to social, emotional and physical factors. Community support, physical care and activity, as well as distancing from work have been found to be particularly efficient. Similarities among burnout strategies include cultivating community and building a sense of shared understanding. Additionally, improving self-awareness and regulating emotions are often the desired outcome of these strategies. Extending these strategies outside of workplace initiatives and into convenient, personal spaces has been suggested to preserve work-life balance.

Thus, narrative medicine offers a space for these strategies to culminate in flash writing. Narrative medicine has been proposed as a model for humane and effective medicine, combining narrative competence and medical practice. Using this model, gaining narrative competence has the ability to positively impact the lives of healthcare professionals and patients, as well as interprofessional teams and broader organizations. The efficacy of flash writing to gain this competence as well as manage the burnout stressors that would typically detract from narrative medicine warrants research into this area.

Flash writing offers the opportunity to investigate the relationship between reflective/ creative writing and burnout. Flash writing can be understood as short-form, creative pieces written in one's personal style. This type of writing exercise can be performed prompted or unprompted, takes approximately 5-10 minutes to complete and is meant to serve the psychological needs of the author. As such, its implementation in burnout alleviation or prevention as well as acute stress reduction may serve as an easily accessible, efficient and customizable strategy.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must be current faculty at Atrium Health Wake Forest Baptist (AHWFB) within three departments: internal medicine, surgery and pediatrics

Exclusion Criteria:

* Faculty who are not currently working at AHWFB may be excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Maslach Burnout Inventory - Human Services Survey (MBI-HSS) | Month 6
  Maslach Burnout Inventory - Human Services Survey, is a questionnaire used to assess burnout among professionals in human service fields. It measures three core dimensions of burnout: Emotional Exhaustion (EE), Depersonalization (DP), and Personal Accomplishment (PA). Each dimension is scored based on the responses to a series of questions, using a 7-point scale (0-6) where higher scores generally indicate higher levels of burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Cormac O'Donovan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No